CLINICAL TRIAL: NCT02387918
Title: Vomiting After Tonsillectomy in Children: A Comparison of Dexamethasone and Acupuncture
Brief Title: Prevention of POV After Paediatric Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohamed Moeen Ibrahim, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SM2015
Record Dates: First submitted 2015-02-27; First posted 2015-03-13 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Vomiting
Keywords: Tonsillectomy; postoperative vomiting (POV); Dexamethasone; Acupuncture
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Patients will receive Intravenous dexamethasone 0.15 mg/kg immediately after induction of anesthesia.
  Interventions: Drug: Dexamethasone
- Acupuncture (Active Comparator): Acupuncture at point Neiguan (Pericardium-6) bilaterally and at point CV13 (Shang Wen) with acupuncture needles (0.25x25 mm) to a depth of approximately 7 mm will be performed on the children immediately after induction of anaesthesia and removed after 20 minutes
  Interventions: Device: Acupuncture

INTERVENTIONS:
Drug: Dexamethasone — Patients will receive Intravenous dexamethasone 0.15 mg/kg immediately after induction of anesthesia.
  Arms: Dexamethasone
Device: Acupuncture — Acupuncture treatment (just after induction of anaesthesia and for approximately 20 minutes)
  Arms: Acupuncture

SUMMARY:
Tonsillectomy is one of the most frequently performed surgical procedures in children. It remains associated with a high morbidity related to postoperative vomiting (POV), pain, risk of bleeding, and dehydration due to impaired oral intake. Current medications for POV have limited efficacy and may even be associated with potential side-effects. Non-pharmacological techniques such as acupuncture has been investigated as alternatives to antiemetics and as additional treatment modalities for POV.

DETAILED DESCRIPTION:
Postoperative vomiting (POV) is one of the most common complication in children undergoing tonsillectomy. Its incidence is between 62% and 73% when no prophylactic antiemetic is given. Because of Limited efficacy and side effects with antiemetics, many alternative treatment had been used. Acupuncture is simple, inexpensive, and noninvasive with minimal side effects. The objective of this study is to compare two prophylactic antiemetic treatments :

* Dexamethasone (0.15 mg/kg) immediately after induction of anaesthesia
* Acupuncture treatment (immediately after induction of anaesthesia and for approximately 20 minutes)

ELIGIBILITY:
Inclusion Criteria:

* children aged 2-8 y.
* children ASA 1-2
* tonsillectomy with or without adenoidectomy

Exclusion Criteria:

* American Society of Anesthesiologists grade greater than or equal to III (patient with severe systemic disease)
* intravenous induction
* contraindication to steroids
* Rash or local infection over an acupuncture point
* administration of steroids in the 24 hours before the surgery
* Use of medication with antiemetic effect within the 24 hours before surgery
* Gastric or intestinal diseases
* refusal of parents

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of POV after tonsillectomy with or without adenoidectomy | 24 hours postoperatively
  by 3 point ordinal scale

CONTACTS AND LOCATIONS:
Overall Officials: Seham Ibrahim, Lecturer, Principal Investigator — health,Higher education
Locations (1):
- Faculty of Medicine Assuit University, Egypt, Assuit, Egypt